CLINICAL TRIAL: NCT05438576
Title: Screening for Peripartum Cardiomyopathies Using Artificial Intelligence (SPEC-AI) in Nigeria
Brief Title: Screening for Pregnancy Related Heart Failure in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Demilade A. Adedinsewo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-000539; K12AR084222 (NIH); UL1TR002377 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Cardiomyopathy; Pregnancy Related
Keywords: Cardiomyopathy; Artificial Intelligence; Women's Health; Digital Health
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will have ECGs analyzed with artificial intelligence for cardiomyopathy detection.
  Interventions: Other: Digital stethoscope electrocardiogram
- Control (No Intervention): Participants will have standard clinical ECGs acquired.

INTERVENTIONS:
Other: Digital stethoscope electrocardiogram — Digital stethoscope artificial intelligence enabled electrocardiogram (AI-ECG). An artificial intelligence algorithm which analyses ECG data and generates prediction probabilities for a diagnosis of cardiomyopathy.
  Arms: Intervention

SUMMARY:
This study will evaluate the effectiveness of an artificial intelligence-enabled ECG (AI-ECG) for cardiomyopathy detection in an obstetric population in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or within 12 months postpartum
* Willing and able to provide informed consent

Exclusion Criteria:

* Complex congenital heart disease (single ventricle physiology or significant shunts with cardiac structural changes)
* Significant conduction abnormalities (ventricular pacing on recorded ECG, pacemaker dependence, or severely abnormal/bizarre QRS morphology on ECG tracings)
* Unable or unwilling to provide consent

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1232 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demilade Adedinsewo, MD, MPH, Principal Investigator — Mayo Clinic
Locations (6):
- Nigeria (6):
  - Rasheed Shekoni Specialist Hospital, Dutse, Jigawa State
  - University of Ilorin Teaching Hospital, Ilorin, Kwara State
  - Olabisi Onabanjo University Teaching Hospital, Sagamu, Ogun State
  - University College Hospital, Ibadan, Oyo State
  - Aminu Kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adedinsewo DA, Morales-Lara AC, Dugan J, Garzon-Siatoya WT, Yao X, Johnson PW, Douglass EJ, Attia ZI, Phillips SD, Yamani MH, Tobah YB, Rose CH, Sharpe EE, Lopez-Jimenez F, Friedman PA, Noseworthy PA, Carter RE. Screening for peripartum cardiomyopathies using artificial intelligence in Nigeria (SPEC-AI Nigeria): Clinical trial rationale and design. Am Heart J. 2023 Jul;261:64-74. doi: 10.1016/j.ahj.2023.03.008. Epub 2023 Mar 25. PMID 36966922
- [Result] Adedinsewo DA, Morales-Lara AC, Afolabi BB, Kushimo OA, Mbakwem AC, Ibiyemi KF, Ogunmodede JA, Raji HO, Ringim SH, Habib AA, Hamza SM, Ogah OS, Obajimi G, Saanu OO, Jagun OE, Inofomoh FO, Adeolu T, Karaye KM, Gaya SA, Alfa I, Yohanna C, Venkatachalam KL, Dugan J, Yao X, Sledge HJ, Johnson PW, Wieczorek MA, Attia ZI, Phillips SD, Yamani MH, Tobah YB, Rose CH, Sharpe EE, Lopez-Jimenez F, Friedman PA, Noseworthy PA, Carter RE; SPEC-AI Nigeria Investigators. Artificial intelligence guided screening for cardiomyopathies in an obstetric population: a pragmatic randomized clinical trial. Nat Med. 2024 Oct;30(10):2897-2906. doi: 10.1038/s41591-024-03243-9. Epub 2024 Sep 2. PMID 39223284

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants had ECGs analyzed with artificial intelligence for cardiomyopathy detection.
  Digital stethoscope electrocardiogram: Digital stethoscope artificial intelligence enabled electrocardiogram (AI-ECG). An artificial intelligence algorithm which analyses ECG data and generates prediction probabilities for a diagnosis of cardiomyopathy.
- Control: Participants had standard clinical ECGs acquired.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 616 | 616
Completed | 587 | 608
Not Completed | 29 | 8
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Not Eligible | 2 | 1
Not completed — Did not complete baseline testing | 22 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 587 | 608 | 1195
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [27 to 35] | 31 [26 to 35] | 31 [27 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 587 | 608 | 1195
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 587 | 608 | 1195
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity - Hausa | 163 | 174 | 337
  Ethnicity - Igbo | 61 | 68 | 129
  Ethnicity - other | 35 | 41 | 76
  Ethnicity - Yoruba | 328 | 325 | 653
Region of Enrollment [Number; unit: participants]
  Nigeria | 587 | 608 | 1195

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF) <50%
Description: Number of participants diagnosed with left ventricular ejection fraction (LVEF) <50% by echocardiography during pregnancy or within 12 months postpartum.
Time Frame: 18 months
Population: Analysis was categorized by pregnant and post-partum participants. Total of each group equals the overall number of participants analyzed per arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 587 | 608
Participants
  Pregnant: number analyzed (Participants) | 423 | 451
  Pregnant | 3 | 1
  Post partum: number analyzed (Participants) | 164 | 157
  Post partum | 21 | 11
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.05 to 4.27]

2. Secondary Outcome: Effectiveness of AI-ECG for Cardiomyopathy Detection in the Intervention Arm for Left Ventricular Ejection Fraction (LVEF) ≤ 35%
Description: This is defined as a positive point-of-care AI prediction for LVEF ≤ 35% (maximum prediction across all stethoscope recording locations) confirmed with echocardiography
Time Frame: 18 months
Population: To explain the differences in number analyzed for each section below, details are provided: Sensitivity, is calculated as True Positive (TP) / (TP + FN), as such the denominator in this case is 17. Specificity is calculated as True Negatives (TN) divided by True Negatives and False Positives (TN + FP), and the denominator is 563. Positive Predictive Value (PPV) = TP / (TP + FP), with a denominator of 122 and Negative Predictive Value (PPV) = TN / (TN + FN) with a denominator of 458.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 587
Participants
  LVEF ≤ 35% (Sensitivity): number analyzed (Participants) | 17
  LVEF ≤ 35% (Sensitivity) | 17
  LVEF ≤ 35% (Specificity): number analyzed (Participants) | 563
  LVEF ≤ 35% (Specificity) | 458
  LVEF ≤ 35% (PPV): number analyzed (Participants) | 122
  LVEF ≤ 35% (PPV) | 17
  LVEF ≤ 35% (NPV): number analyzed (Participants) | 458
  LVEF ≤ 35% (NPV) | 458

3. Secondary Outcome: Effectiveness AI-ECG for Cardiomyopathy Detection in the Intervention Arm in LVEF < 40%
Description: This is defined as a positive point-of-care AI prediction for LVEF < 40% (maximum prediction across all stethoscope recording locations) confirmed with echocardiography
Time Frame: 18 months
Population: To explain the differences in number analyzed for each section below, details are provided: Sensitivity, is calculated as True Positive (TP) / (TP + FN), as such the denominator in this case is 20. Specificity is calculated as True Negatives (TN) divided by True Negatives and False Positives (TN + FP), and the denominator is 560. Positive Predictive Value (PPV) = TP / (TP + FP), with a denominator of 122 and Negative Predictive Value (PPV) = TN / (TN + FN) with a denominator of 458.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 587
Participants
  LVEF < 40% (Sensitivity): number analyzed (Participants) | 20
  LVEF < 40% (Sensitivity) | 20
  LVEF < 40% (Specificity): number analyzed (Participants) | 560
  LVEF < 40% (Specificity) | 458
  LVEF < 40% (PPV): number analyzed (Participants) | 122
  LVEF < 40% (PPV) | 20
  LVEF < 40% (NPV): number analyzed (Participants) | 458
  LVEF < 40% (NPV) | 458

4. Secondary Outcome: Effectiveness AI-ECG for Cardiomyopathy Detection in the Intervention Arm in LVEF < 45%
Description: This is defined as a positive point-of-care AI prediction for LVEF <45% (maximum prediction across all stethoscope recording locations) confirmed with echocardiography
Time Frame: 18 months
Population: To explain the differences in number analyzed for each section below, details are provided: Sensitivity, is calculated as True Positive (TP) / (TP + FN), as such the denominator in this case is 23. Specificity is calculated as True Negatives (TN) divided by True Negatives and False Positives (TN + FP), and the denominator is 557. Positive Predictive Value (PPV) = TP / (TP + FP), with a denominator of 122 and Negative Predictive Value (PPV) = TN / (TN + FN) with a denominator of 458.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 587
Participants
  LVEF < 45% (Sensitivity): number analyzed (Participants) | 23
  LVEF < 45% (Sensitivity) | 22
  LVEF < 45% (Specificity): number analyzed (Participants) | 557
  LVEF < 45% (Specificity) | 457
  LVEF < 45% (PPV): number analyzed (Participants) | 122
  LVEF < 45% (PPV) | 22
  LVEF < 45% (NPV): number analyzed (Participants) | 458
  LVEF < 45% (NPV) | 457

5. Secondary Outcome: Effectiveness AI-ECG for Cardiomyopathy Detection in the Intervention Arm in LVEF < 50%
Description: This is defined as a positive point-of-care AI prediction for LVEF <50% (maximum prediction across all stethoscope recording locations) confirmed with echocardiography
Time Frame: 18 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 587
Participants
  LVEF < 50% (Sensitivity): number analyzed (Participants) | 23
  LVEF < 50% (Sensitivity) | 22
  LVEF < 50% (Specificity): number analyzed (Participants) | 557
  LVEF < 50% (Specificity) | 457
  LVEF < 50% (PPV): number analyzed (Participants) | 122
  LVEF < 50% (PPV) | 22
  LVEF < 50% (NPV): number analyzed (Participants) | 458
  LVEF < 50% (NPV) | 457

6. Other Pre Specified Outcome: Composite Adverse Cardiovascular Events
Description: The number of subjects to experience composite cardiovascular events with include any of the following: diastolic heart failure, gestational hypertension, pre-eclampsia, eclampsia, valvular heart disease, atrial arrhythmias and sustained ventricular arrhythmias.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 587 | 608
Participants | 56 | 53
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.621, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.74 to 1.64]

7. Other Pre Specified Outcome: Echocardiography Utilization
Description: Determine the impact of an AI-ECG on echocardiography utilization
Time Frame: 18 months
Population: Data was not collected nor analyzed for this outcome measure
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Effectiveness of AI Point of Care Tools for Cardiomyopathy Detection in the Intervention Arm
Description: Develop and evaluate the diagnostic performance of an AI-enhanced point of care screening tool
Time Frame: 18 months
Population: Data was not collected nor analyzed for this outcome measure
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Long-term clinical outcomes including mortality were passively tracked for all participants (for up to 18 months) beyond the duration of active trial participation. These outcomes are also described as "adverse cardiovascular events" in order to match prevailing descriptions in published literature but are completely unrelated to the study intervention. Study defined adverse events per protocol were collected for up to 3 hours following study intervention (ECG and Echo recording).
Description: Anticipated study related risk is limited to potential skin irritation from placement of ECG lead electrode stickers directly on the skin for ECG measurements. The "adverse cardiovascular events" reported in the manuscript are not "events" in the context of this clinical trial. They are described collectively as "adverse cardiovascular events" to facilitate a comprehensive grouping for descriptive and summarization purposes, and to ensure consistency with the existing literature.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 12/587 | 3/608
Serious Adverse Events (participants affected / at risk) | 56/587 | 53/608
Other Adverse Events (participants affected / at risk) | 1/587 | 4/608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=587) | Control (N=608)
Diastolic heart failure (Cardiac disorders) | 2 | 1 — Non-treatment related (not related to study intervention)
Atrial Arrhythmias (Cardiac disorders) | 0 | 0 — Non-treatment related (not related to study intervention)
Sustained Ventricular Arrhythmias (Cardiac disorders) | 0 | 0 — Non-treatment related (not related to study intervention)
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 30 | 30 — Non-treatment related (not related to study intervention)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 21 | 19 — Non-treatment related (not related to study intervention)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 6 | 4 — Non-treatment related (not related to study intervention)
Valvular Disease (Cardiac disorders) | 1 | 1 — Non-treatment related (not related to study intervention)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=587) | Control (N=608)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT05438576/Prot_SAP_000.pdf